CLINICAL TRIAL: NCT06919198
Title: Procedural Sedation for Minor Procedures Using Jet-Injected Subcutaneous Ketamine
Brief Title: The Dreamy Jet Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: IND application was not approved
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1429; A536750 (Other: UW Madison); SMPH\PEDIATRICS\PICU (Other: UW Madison); Protocol Version 12/20/24 (Other: UW Madison)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Sedation; Blood Drawing Procedure; Immunization; IV Placement
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- J-tip jet injection (Experimental): Participants will be given ketamine via J-tip jet injection
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — ketamine 2.5 mg/kg

SUMMARY:
The goal of this clinical trial is to see if a device known as a jet-injection system can help deliver a single dose of a sedating medication with less pain and stress than current methods.

Participants will receive a dose of the sedative in their arm or thigh before their procedure at the sedation clinic.

DETAILED DESCRIPTION:
This study will evaluate whether jet-injected ketamine can provide adequate sedation to perform minimally invasive procedures in children with heightened procedural sensitivity in a pediatric sedation clinic environment. Minimally invasive procedures include, but are not limited to, blood draws, IV placement, and immunizations.

ELIGIBILITY:
Inclusion Criteria:

* Referred to UW Health American Family Children's Hospital Pediatric Sedation Clinic for minimally invasive procedures such as blood draw, IV placement, or immunization
* Age 2-15 years
* Weight <40kg

Exclusion Criteria:

* Participants with elevated intracranial pressure
* Participants with uncontrolled hypertension
* Participants who are pregnant or possibly pregnant (i.e., people of child bearing potential unable to provide a negative pregnancy test)
* Participants who received a dose of medication within 2 hours of their appointment with the intention of sedation (i.e., benzodiazepines, opioids, alpha-2 agonists, 1st generation antihistamines)
* Participants who are receiving medications which might enhance the sympathomimetic effect of ketamine (i.e., theophylline, aminophylline, amphetamine, or pseudoephedrine)
* Participants who are receiving medications that might interfere with the expected pharmacokinetics of ketamine (i.e., ketoconazole, clarithromycin, rifampin, or carbamazepine)
* Participant's parent/legal guardian requires a translator for communication about the patient's medical care

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of procedural success | Up to 3 hours
  Feasibility is measured by completion of the procedure using only the study drug. It is indicated by "yes" or "no".

SECONDARY OUTCOMES:
Rate of procedural success | Up to 3 hours
  Percentage of participants who are able to complete the procedure using only the study intervention.
Time it takes to achieve target PSSS score | Up to 20 minutes
  Time to PSSS score is measured from time of injection until target PSSS is achieved.
Rate of adverse events | Up to 3 hours
  Reported as a percentage of total participants who experience an adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Peters, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No